CLINICAL TRIAL: NCT01177722
Title: Lot-to-Lot Consistency Study of DTaP-IPV-Hep B-PRP-T Vaccine Administered at 2-4-6 Months of Age in Healthy Latin American Infants Concomitantly With Prevenar™ and Rotarix™
Brief Title: A Study of DTaP-IPV-Hep B-PRP-T Vaccine Given With Prevenar™ and Rotarix™ in Healthy Latin American Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A3L24; UTN: U1111-1111-5801 (Other: WHO)
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis
Keywords: Diphtheria; Tetanus; Whooping cough; Hepatitis B; Poliomyelitis; Diphtheria-Tetanus-acellular Pertussis Vaccines
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: DTaP-IPV-Hep B-PRP-T (Lot A) (Experimental)
  Interventions: Biological: DTaP-IPV-Hep B-PRP-T Vaccine
- Group 2: DTaP-IPV-Hep B-PRP-T (Lot B) (Experimental)
  Interventions: Biological: DTaP-IPV-Hep B-PRP-T Vaccine
- Group 3: DTaP-IPV-Hep B-PRP-T (Lot C) (Experimental)
  Interventions: Biological: DTaP-IPV-Hep B-PRP-T Vaccine
- Group 4: Active Control (Active Comparator)
  Interventions: Biological: DTaP-Hep B-IPV vaccine

INTERVENTIONS:
Biological: DTaP-IPV-Hep B-PRP-T Vaccine — 0.5 mL, Intramuscular
  Arms: Group 1: DTaP-IPV-Hep B-PRP-T (Lot A)
Biological: DTaP-IPV-Hep B-PRP-T Vaccine — 0.5 mL, Intramuscular
  Arms: Group 2: DTaP-IPV-Hep B-PRP-T (Lot B)
Biological: DTaP-IPV-Hep B-PRP-T Vaccine — 0.5 mL, Intramuscular
  Arms: Group 3: DTaP-IPV-Hep B-PRP-T (Lot C)
Biological: DTaP-Hep B-IPV vaccine — 0.5 mL, Intramuscular
  Other Names: Infanrix hexa™
  Arms: Group 4: Active Control

SUMMARY:
The purpose of this study is to generate immunogenicity and safety data of an investigational hexavalent DTaP-IPV-Hep B-PRP-T vaccine compared to a control vaccine, Infanrix hexa™ when given along with Prevenar™ and Rotarix™ vaccines.

Primary Objectives:

* To demonstrate the equivalence of immunogenicity of 3 lots of DTaP-IPV-Hep B-PRP-T vaccine 1 month after a 3-dose primary series (2, 4 and 6 months) when given with Prevenar™ and Rotarix™, in terms of immunoresponses.
* To demonstrate the non-inferiority of the hexavalent DTaP-IPV-Hep B-PRP-T vaccine to the licensed hexavalent Infanrix hexa vaccine when given with Prevenar™ and Rotarix™.

Secondary Objectives:

* To describe in each group the immunogenicity parameters for all antigens for each vaccine
* To assess the safety profile in terms of solicited and unsolicited adverse events and serious adverse events in each group for each vaccine.

DETAILED DESCRIPTION:
Each participant will receive 3 doses of 1 of 3 lots of the investigational hexavalent vaccine or the control vaccine, Infanrix hexa™, administered with Prevenar™ at 2, 4, and 6 months of age and Rotarix™ at 2 and 4 months of age.

All participants will be monitored for safety for 6 months after the last injection of the primary vaccination series.

ELIGIBILITY:
Inclusion Criteria :

* Two month old infants (55 to 65 days old) on the day of inclusion.
* Born at full term of pregnancy (≥ 37 weeks) with a birth weight ≥ 2.5 kg.
* Informed consent form signed by one or both parents or by the legally acceptable representative as per local requirements.
* Able to attend all scheduled visits and to comply with all trial procedures.
* Received Hepatitis B and Bacille de Calmette-Guérin (BCG) vaccines between birth and one month of life in agreement with the national immunization calendar.

Exclusion Criteria :

* Participation in another clinical trial in the 4 weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy, or long-term systemic corticosteroid therapy.
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances.
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator.
* Blood or blood-derived products received since birth that might interfere with the assessment of the immune response.
* Any vaccination before trial vaccination (except Hepatitis B and Bacille de Calmette Guérin given at birth).
* Any planned vaccination until 1 month after the last trial vaccination (except the study vaccines, rotavirus and pneumococcal conjugated vaccines).
* Documented history of pertussis, tetanus, diphtheria, poliomyelitis, Haemophilus influenzae type b or Hepatitis B infection(s) (confirmed either clinically, serologically or microbiologically).
* Previous vaccination against pertussis, tetanus, diphtheria, poliomyelitis, or Haemophilus influenzae type b infections.
* Known personal or maternal history of Human Immunodeficiency Virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C seropositivity.
* Known coagulopathy, thrombocytopenia or a bleeding disorder preceding inclusion contraindicating intramuscular (IM) vaccination.
* History of seizures or encephalopathy.
* Febrile illness (temperature ≥ 38.0°C), or moderate or severe acute illness/infection on the day of inclusion, according to the Investigator judgment.

Ages: 55 Days to 65 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1375 (Actual)
Dates: Start 2010-08; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Cali, Colombia
- San José, Costa Rica

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 03 August 2010 to 23 November 2010 in 2 clinical centers in Columbia and 1 clinical center in Costa Rica.
Pre-assignment Details: A total of 1375 participants who met all inclusion criteria and none of the exclusion criteria were enrolled and vaccinated.
Groups:
- DTap-IPV-Hep B-PRP~T Batch A: Participants received a 3-dose primary series of vaccinations with Batch A of diphtheria, tetanus, pertussis (2-component acellular), recombinant hepatitis B (Hep B) Hansenula polymorpha and poliomyelitis vaccine adsorbed, and Haemophilus influenzae type b (Hib) vaccine [polyribosyl ribitol phosphate (PRP) conjugated to tetanus protein (DTaP-IPV-Hep B-PRP~T), with one dose each at 2, 4, and 6 months of age. Prevenar™ was co-administered with study vaccine at 2, 4, and 6 months of age, and Rotarix™ was co-administered at 2 and 4 months of age.
- DTaP-IPV-Hep B-PRP~T Batch B: Participants received a 3-dose primary series of vaccinations with Batch B of diphtheria, tetanus, pertussis (2-component acellular), recombinant hepatitis B (Hep B) Hansenula polymorpha and poliomyelitis vaccine adsorbed, and Haemophilus influenzae type b (Hib) vaccine [polyribosyl ribitol phosphate (PRP) conjugated to tetanus protein (DTaP-IPV-Hep B-PRP~T), with one dose each at 2, 4, and 6 months of age. Prevenar™ was co-administered with study vaccine at 2, 4, and 6 months of age, and Rotarix™ was co-administered at 2 and 4 months of age.
- DTaP-IPV-Hep B-PRP~T Batch C: Participants received a 3-dose primary series of vaccinations with Batch C of diphtheria, tetanus, pertussis (2-component acellular), recombinant hepatitis B (Hep B) Hansenula polymorpha and poliomyelitis vaccine adsorbed, and Haemophilus influenzae type b (Hib) vaccine [polyribosyl ribitol phosphate (PRP) conjugated to tetanus protein (DTaP-IPV-Hep B-PRP~T), with one dose each at 2, 4, and 6 months of age. Prevenar™ was co-administered with study vaccine at 2, 4, and 6 months of age, and Rotarix™ was co-administered at 2 and 4 months of age.
- Infanrix Hexa: Participants received a 3-dose primary series of vaccinations with the licensed Infanrix hexa™, with one dose each at 2, 4, and 6 months of age. Prevenar™ was co-administered with study vaccine at 2, 4, and 6 months of age, and Rotarix™ was co-administered at 2 and 4 months of age.
Period: Overall Study
Arm/Group | DTap-IPV-Hep B-PRP~T Batch A | DTaP-IPV-Hep B-PRP~T Batch B | DTaP-IPV-Hep B-PRP~T Batch C | Infanrix Hexa
Started | 344 (A Batch B participant got Batch A vaccine data analyses was according to actual vaccine administered) | 344 (A randomized participant got Batch A vaccine, analyses was according to actual vaccine administered.) | 342 | 345
Completed | 331 | 334 | 333 | 338
Not Completed | 13 | 10 | 9 | 7
Not completed — Serious Adverse Event | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 4 | 3 | 1
Not completed — Withdrawal by Subject | 10 | 6 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTap-IPV-Hep B-PRP~T Batch A | DTaP-IPV-Hep B-PRP~T Batch B | DTaP-IPV-Hep B-PRP~T Batch C | Infanrix Hexa | Total
Number analyzed (Participants) | 344 | 344 | 342 | 345 | 1375
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 344 | 344 | 342 | 345 | 1375
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] | 58.8 (3.49) | 58.7 (3.25) | 58.5 (3.16) | 58.7 (3.31) | 58.7 (3.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 165 | 152 | 156 | 634
  Male | 183 | 179 | 190 | 189 | 741
Region of Enrollment [Number; unit: Participants]
  Colombia | 233 | 234 | 233 | 233 | 933
  Costa Rica | 111 | 110 | 109 | 112 | 442

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Anti-Hepatitis B Before and After 3 Dose Primary Vaccination With Either DTaP-IPV-Hep B-PRP~T Batch A, B, or C, or Infanrix Hexa™
Description: Antibodies against Hepatitis B (Hep B) were measured by chemiluminescence detection.
Time Frame: Day 0 (pre-vaccination) Dose 1 and 30 days post-vaccination
Population: GMTs were assessed in all subjects who did not have any protocol violation that might interfere with primary criteria evaluation (Per-Protocol Population).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | DTap-IPV-Hep B-PRP~T Batch A | DTaP-IPV-Hep B-PRP~T Batch B | DTaP-IPV-Hep B-PRP~T Batch C | Infanrix Hexa
Number analyzed (Participants) | 312 | 310 | 313 | 316
Titers
  Anti-Hep B Pre-dose 1 | 4.02 [3.50 to 4.61] | 4.07 [3.58 to 4.62] | 4.93 [4.20 to 5.79] | 4.30 [3.68 to 5.03]
  Anti-Hep B Post-dose 3 | 3048 [2672 to 3476] | 2801 [2467 to 3181] | 3202 [2794 to 3668] | 2766 [2466 to 3102]

2. Primary Outcome: Number of Participants With Seroprotection or Vaccine Response After Vaccination With Either DTaP-IPV-Hep B-PRP~T or Infanrix Hexa Vaccine
Description: Seroprotection was defined as titers ≥ 0.01 IU/mL for Diphtheria (D) and Tetanus (T); ≥ 10 IU/mL for Hep B; ≥ 0.15 µg/mL for PRP, and ≥ 8 (1/dil) for Poliovirus. Vaccine response for PT and FHA were defined as a titer ≥ lower limit of quantitation (LLOQ) in initially seronegative participants, or at least persistence (post-vaccination titer ≥ pre-vaccination titer) in initially seropositive subjects (titer ≥ LLOQ).
Time Frame: 30 Days post-dose 3
Population: Seroprotection and vaccine response were assessed in all subjects who did not have any protocol violation that might interfere with primary criteria evaluation (Per Protocol Population).
Measure: Number; unit: Participants
Arm/Group | DTap-IPV-Hep B-PRP~T Batch A | DTaP-IPV-Hep B-PRP~T Batch B | DTaP-IPV-Hep B-PRP~T Batch C | Infanrix Hexa
Number analyzed (Participants) | 312 | 310 | 313 | 316
Participants
  Anti-Diphtheria (N = 310, 310, 312, 315) | 310 | 310 | 312 | 315
  Anti-Tetanus (N = 311, 310, 311, 314) | 311 | 310 | 311 | 314
  Anti-PT (N = 308, 309, 308, 312) | 304 | 299 | 299 | 307
  Anti-FHA (N = 306, 306, 304, 311) | 306 | 305 | 303 | 309
  Anti-Polio 1 (N = 310, 309, 308, 311) | 310 | 309 | 308 | 311
  Anti-Polio 2 (N = 309, 309, 307, 312) | 309 | 309 | 307 | 312
  Anti-Polio 3 (N = 310, 309, 307, 312) | 310 | 309 | 307 | 311
  Anti-Hep B (N = 312, 310, 312, 316) | 311 | 310 | 310 | 316
  Anti-PRP (N = 312, 310, 312, 316) | 299 | 298 | 287 | 303

3. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies After Vaccination With Either DTaP-IPV-Hep B-PRP~T or Infanrix Hexa Vaccine
Description: Antibodies were measured by toxin neutralization test for Diphtheria (D); enzyme-linked immunosorbent assay (ELISA) for Tetanus (T), Pertussis toxoid (PT), and Filamentous hemagglutinin (FHA); neutralization assay for Poliovirus types 1, 2, and 3; chemiluminescence detection for Hepatitis B (Hep B), and Farr type radioimmunoassay for Haemophilus influenza type b (PRP).
Time Frame: Day 0 (pre-vaccination) and 30 days post-dose 3
Population: GMTs were assessed in all subjects who did not have any protocol violation that might interfere with primary criteria evaluation (Per Protocol Population).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Infanrix Hexa™: Participants received a 3-dose primary series of vaccinations with the licensed Infanrix hexa™, with one dose each at 2, 4, and 6 months of age. Prevenar™ was co-administered with study vaccine at 2, 4, and 6 months of age, and Rotarix™ was co-administered at 2 and 4 months of age.
Arm/Group | DTap-IPV-Hep B-PRP~T Batch A | DTaP-IPV-Hep B-PRP~T Batch B | DTaP-IPV-Hep B-PRP~T Batch C | Infanrix Hexa™
Number analyzed (Participants) | 312 | 310 | 313 | 316
Titers
  Anti-Diphtheria Pre-dose 1 (N= 312, 308, 311, 315) | 0.599 [0.513 to 0.699] | 0.596 [0.505 to 0.703] | 0.641 [0.547 to 0.752] | 0.630 [0.530 to 0.749]
  Anti-Diphtheria Post-dose 3 (N=310, 310, 312, 315) | 0.252 [0.224 to 0.285] | 0.279 [0.247 to 0.316] | 0.228 [0.201 to 0.260] | 0.240 [0.214 to 0.269]
  Anti-Tetanus Post-dose 3 (N = 311, 310, 311, 314) | 1.66 [1.54 to 1.78] | 1.55 [1.43 to 1.68] | 1.45 [1.33 to 1.59] | 1.80 [1.69 to 1.93]
  Anti-PT Pre-dose 1 (N = 308, 309, 310, 314) | 3.02 [2.65 to 3.45] | 3.50 [3.03 to 4.04] | 3.54 [3.10 to 4.05] | 3.11 [2.70 to 3.59]
  Anti-PT Post-dose 3 (N = 312, 310, 311, 314) | 102 [96.1 to 108] | 103 [95.9 to 110] | 102 [95.0 to 110] | 98.9 [92.3 to 106]
  Anti-FHA Pre-dose 1(N = 307, 307, 307, 312) | 5.36 [4.77 to 6.02] | 5.66 [5.01 to 6.39] | 5.76 [5.12 to 6.49] | 5.13 [4.61 to 5.70]
  Anti-FHA Post-dose 3 (N=311, 309, 310, 315) | 186 [174 to 199] | 175 [163 to 188] | 183 [171 to 197] | 118 [110 to 127]
  Anti-Polio 1 Post-dose 3 (N = 310, 309, 308, 311) | 755 [674 to 847] | 655 [580 to 739] | 636 [561 to 722] | 1298 [1151 to 1464]
  Anti-Polio 2 Post-dose 3 (N = 309, 309, 307, 312) | 1190 [1054 to 1344] | 1232 [1101 to 1379] | 1120 [994 to 1261] | 1981 [1756 to 2234]
  Anti-Polio 3 Post-dose 3 (N = 310, 309, 307, 312) | 1102 [972 to 1250] | 1119 [975 to 1284] | 1097 [963 to 1250] | 1944 [1680 to 2249]
  Anti-PRP Post-dose 3 (N = 312, 310, 312, 316) | 3.37 [2.80 to 4.05] | 4.02 [3.35 to 4.82] | 3.33 [2.72 to 4.07] | 2.24 [1.90 to 2.64]

4. Secondary Outcome: Number of Participants Reporting at Least One Solicited Injection Site (Study Vaccine) or Systemic Reactions After Vaccination With Either DTaP-IPV-Hep B-PRP~T or Infanrix Hexa Vaccine
Description: Solicited Injection Site Reactions: Pain, Erythema, and Swelling. Solicited Systemic Reactions: Pyrexia (Temperature), Vomiting, Crying, Somnolence, Anorexia,and Irritability. Grade 3 was defined as: Pain, cries when injected limb is moved or movement of the limb is reduced; Erythema and Swelling, ≥ 5 cm; Pyrexia, (Temperature) ≥ 39.6°C; Vomiting, ≥ 6 episodes/24 hours or requiring parenteral hydration; Crying, > 3 hours; Somnolence, sleeping most of time or difficult to wake up; Anorexia, refuses ≥ 3 feed/meals or refuses most feeds/meals; and Irritability, inconsolable.
Time Frame: Day 0 up to 7 after each dose
Population: Solicited injection site and systemic reactions were assessed in all participants who received at least one dose of study vaccine (Safety Analysis Set).
Measure: Number; unit: Participants
Arm/Group | DTap-IPV-Hep B-PRP~T Batch A | DTaP-IPV-Hep B-PRP~T Batch B | DTaP-IPV-Hep B-PRP~T Batch C | Infanrix Hexa
Number analyzed (Participants) | 345 | 343 | 342 | 345
Participants
  Pain Post-dose 1 (N = 338, 341, 340, 344) | 199 | 194 | 216 | 185
  Pain Post-dose 2 (N = 333, 337, 335, 340) | 180 | 196 | 203 | 188
  Pain Post-dose 3 (N = 331, 331, 334, 337) | 168 | 163 | 162 | 147
  Grade 3 Pain Post Dose 1 (N = 338, 341, 344, 344) | 21 | 22 | 22 | 7
  Grade 3 Pain Post Dose 3 (N=331, 331, 334, 338) | 10 | 9 [0 to 0] | 8 | 8
  Erythema Post-dose 1 (N = 338, 341, 340, 344 | 72 | 63 | 82 | 52
  Erythema Post-dose 2 (N = 333, 337, 335, 340 | 87 | 78 | 80 | 67
  Erythema Post-dose 3 (N = 331, 331, 334, 337) | 85 | 79 | 96 | 68
  Grade 3 Erythema Post-dose 1(N=338, 341, 340, 344) | 2 | 3 | 2 | 0
  Grade 3 Erythema Post-dose 3(N=331, 331, 334, 337) | 0 | 0 | 1 | 0
  Swelling Post dose 1 (N = 338, 341, 340, 344) | 47 | 30 | 47 | 33
  Swelling Post dose 2 (N = 333, 337, 335, 340) | 44 | 35 | 45 | 44
  Swelling Post dose 3 (N = 331, 331, 334, 337) | 43 | 34 | 48 | 42
  Grade 3 Swelling Post-dose 1(N=338, 341, 340, 344) | 2 | 3 | 2 | 0
  Grade 3 Swelling post-dose 3(N=331, 331, 340, 338) | 0 | 0 | 0 | 0
  Pyrexia Post dose 1 (N = 338, 341, 340, 344) | 46 | 42 | 68 | 46
  Pyrexia Post dose 2 (N = 333, 337, 335, 340) | 70 | 68 | 68 | 70
  Pyrexia Post dose 3 (N = 331, 331, 333, 337) | 67 | 63 | 72 | 65
  Grade 3 Pyrexia Post-dose 1 (N=338, 341, 340, 344) | 2 | 0 | 0 | 0
  Grade 3 Pyrexia Post-dose 3 (N=331, 331, 333, 337) | 4 | 1 | 1 | 2
  Vomiting Post dose 1 (N = 338, 341, 340, 344) | 85 | 90 | 86 | 94
  Vomiting Post dose 2 (N = 333, 337, 335, 340) | 58 | 80 | 64 | 62
  Vomiting Post dose 3 (N = 331, 331, 334, 337) | 32 | 58 | 46 | 39
  Grade 3 Vomiting Post-dose 1(N=338, 341, 340, 344) | 4 | 5 | 6 | 5
  Grade 3 Vomiting post-dose 3(N=331, 331, 334, 337) | 3 | 1 | 2 | 2
  Crying Post dose 1 (N = 338, 341, 340, 344) | 198 | 186 | 189 | 161
  Crying Post dose 2 (N = 333, 337, 335, 340) | 163 | 179 | 169 | 161
  Crying Post dose 3 (N = 331, 331, 334, 337) | 141 | 145 | 142 | 120
  Grade 3 Crying Post-dose 1 (N =338, 341, 340, 344) | 15 | 10 | 23 | 9
  Grade 3 Crying Post-dose 3 (N =331, 331, 334, 337) | 8 | 6 | 10 | 6
  Somnolence Post dose 1 (N = 338, 341, 341, 344) | 159 | 146 | 160 | 147
  Somnolence Post dose 2 (N = 333, 337, 335, 340) | 109 | 108 | 110 | 111
  Somnolence Post dose 3 (N = 331, 331, 334, 337) | 85 | 99 | 96 | 81
  Grad 3 Somnolence Post-dose 1 N=338, 341, 341, 344 | 3 | 14 | 19 | 9
  Grad 3 Somnolence Post-dose 3 N=331, 331, 334, 337 | 5 | 2 | 4 | 4
  Anorexia Post dose 1 (N = 338, 341, 341, 344) | 78 | 97 | 96 | 75
  Anorexia Post dose 2 (N = 333, 337, 335, 340) | 75 | 93 | 86 | 74
  Anorexia Post dose 3 (N = 331, 331, 334, 337) | 63 | 64 | 60 | 54
  Grade 3 Anorexia Post-dose 1(N=338, 341, 341, 344) | 3 | 4 | 8 | 3
  Grade 3 Anorexia Post-dose 3(N=331, 331, 334, 337) | 4 | 7 | 4 | 3
  Irritability Post dose 1 (N = 338, 341, 341, 344) | 208 | 206 | 208 | 180
  Irritability Post dose 2 (N = 333, 337, 335, 340) | 193 | 199 | 191 | 193
  Irritability Post dose 3 (N = 331, 332, 334, 337) | 155 | 161 | 154 | 144
  Grd 3 Irritability Post-dose 1N=338, 341, 341, 344 | 15 | 17 | 20 | 8
  Grd 3 Irritability Post-dose 3N=331, 332, 334, 337 | 11 | 13 | 12 | 5

5. Secondary Outcome: Number of Participants Reporting at Least One Solicited Injection Site Reaction at the Prevenar Injection Site After Vaccination With Either DTaP-IPV-Hep B-PRP~T or Infanrix Hexa™ Vaccine
Description: Solicited Injection Site Reactions: Pain, Erythema, and Swelling. Solicited Systemic Reactions: Pyrexia (Temperature), Vomiting, Crying, Somnolence, Anorexia, and Irritability. Grade 3 was defined as: Pain, cries when injected limb is moved or movement of the limb is reduced; Erythema and Swelling, ≥ 5 cm; Pyrexia (Temperature), ≥ 39.6ºC; Vomiting, ≥ 6 episodes/24 hours or requiring parenteral hydration; Crying, > 3 hours; Somnolence, sleeping most of time or difficult to wake up; Anorexia, refuses ≥ 3 feed/meals or refuses most feeds/meals; and Irritability, inconsolable.
Time Frame: Day 0 up to 7 post each vaccination
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | DTap-IPV-Hep B-PRP~T Batch A | DTaP-IPV-Hep B-PRP~T Batch B | DTaP-IPV-Hep B-PRP~T Batch C | Infanrix Hexa
Number analyzed (Participants) | 345 | 341 | 342 | 345
Participants
  Pain Post-dose 1 (N = 338, 341, 340, 344) | 171 | 173 | 184 | 169
  Grade 3 Pain Post-dose 1 (N = 338, 341, 340, 344) | 15 | 15 | 16 | 8
  Pain Post-dose 2 (N = 333, 337, 335, 340) | 160 | 183 | 180 | 174
  Grade 3 Pain Post-dose 2 (N = 333, 337, 335, 340) | 14 | 17 | 16 | 13
  Pain Post-dose 3 (N =331, 331, 334, 337) | 146 | 105 | 146 | 125
  Grade 3 Pain Post-dose 3 (N = 331, 331, 334, 337) | 8 | 9 | 10 | 7
  Erythema Post-dose 1 (N = 338, 341, 340, 344) | 47 | 48 | 55 | 42
  Grade 3 Erythema Post-dose 1 (N=338, 341, 340, 344 | 0 | 1 | 2 | 0
  Erythema Post-dose 2 (N = 333, 337, 335, 340) | 65 | 55 | 62 | 53
  Grade 3 Erythema Post-dose 2 (N=333, 337, 335, 340 | 1 | 0 | 0 | 0
  Erythema Post-dose 3 (N = 331, 331, 334, 337) | 63 | 57 | 69 | 49
  Grade 3 Erythema Post-dose 3 (N=331, 331, 334, 337 | 1 | 1 | 0 | 0
  Swelling Post-dose 1 (N = 338, 341, 340, 344) | 34 | 21 | 33 | 31
  Grade 3 Swelling Post-dose 1 (N=338, 341, 340, 344 | 0 | 0 | 2 | 1
  Swelling Post-dose 2 (N = 333, 337, 335, 340) | 32 | 28 | 36 | 32
  Grade 3 Swelling Post-dose 2 (N=333, 337, 335, 340 | 0 | 0 | 1 | 0
  Swelling Post-dose 3 (N = 331, 331, 334, 337) | 27 | 29 | 36 | 29
  Grade 3 Swelling Post-dose 3 (N=331, 331, 334, 337 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 after Dose 1 through up to 6 months after the last dose.
Description: A participant randomized to Batch B got the Batch A vaccine, safety analyses was according to the actual vaccine administered. Total number reported for each solicited event reflects those with available data for the indicated event.
Arm/Group | DTap-IPV-Hep B-PRP~T Batch A | DTaP-IPV-Hep B-PRP~T Batch B | DTaP-IPV-Hep B-PRP~T Batch C | Infanrix Hexa
Serious Adverse Events (participants affected / at risk) | 10/345 | 14/343 | 16/342 | 10/345
Other Adverse Events (participants affected / at risk) | 208/345 | 206/343 | 216/342 | 193/345
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTap-IPV-Hep B-PRP~T Batch A (N=345) | DTaP-IPV-Hep B-PRP~T Batch B (N=343) | DTaP-IPV-Hep B-PRP~T Batch C (N=342) | Infanrix Hexa (N=345)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral Atrophy Congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sudden Infant Death Syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 5 (5) | 6 (6) | 9 (10) | 8 (8)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dengue Fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Exanthema Subitum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kawasaki's Disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis Media Acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 5 (6) | 11 (11) | 5 (7)
Pneumonia Primary Atypical (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia Viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 2 (3) | 2 (2) | 3 (3)
Viral Diarrhoea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diaphragmatic Hernia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign Body Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DTap-IPV-Hep B-PRP~T Batch A (N=345) | DTaP-IPV-Hep B-PRP~T Batch B (N=343) | DTaP-IPV-Hep B-PRP~T Batch C (N=342) | Infanrix Hexa (N=345)
Vomiting (Gastrointestinal disorders) | 85/338 (85) | 90/341 (90) | 86/340 (86) | 94/344 (94)
Injection Site Erythema (General disorders) | 87/338 (87) | 79/341 (79) | 96/340 (96) | 68/344 (68)
Injection Site Pain (General disorders) | 199/338 (199) | 196/341 (196) | 216/340 (216) | 188/344 (188)
Injection Site Swelling (General disorders) | 47/338 (47) | 35/341 (35) | 48/340 (48) | 44/344 (44)
Irritability (General disorders) | 208/338 (208) | 206/341 (206) | 208/341 (208) | 193/344 (193)
Pyrexia (General disorders) | 70/338 (70) | 68/341 (68) | 72/340 (72) | 70/344 (70)
Nasopharyngitis (Infections and infestations) | 99 (125) | 96 (132) | 90 (116) | 87 (105)
Anorexia (Metabolism and nutrition disorders) | 75/338 (75) | 97/341 (97) | 96/341 (96) | 75/344 (75)
Somnolence (Nervous system disorders) | 159/338 (159) | 146/341 (146) | 160/341 (160) | 147/344 (147)
Crying (Psychiatric disorders) | 198/338 (198) | 186/341 (186) | 189/340 (189) | 161/344 (161)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (24) | 17 (17) | 23 (25) | 17 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.